CLINICAL TRIAL: NCT05455307
Title: Efficacy and Safety of Self-expanding Ureteral Stent for Treating Refractory Ureteral Stricture: Results of a Multicenter Experience
Brief Title: Efficacy and Safety of Allium Ureteral Stent for Treating Refractory Ureteral Stricture
Acronym: Allium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: En Chu Kong Hospital (Other)
Responsible Party: Principal Investigator, ChungChengWang, Chief of department of Urology, En Chu Kong Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eck20200608
Record Dates: First submitted 2022-06-08; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Ureteral Stenosis; Hydronephrosis; Ureteral Stent Occlusion
Keywords: ureteral stone; ureteral stricture; hydronephrosis
MeSH Terms: conditions — Hydronephrosis; Ureterolithiasis

STUDY DESIGN:
Intervention Model Description: single group without control
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental): single arm without placebo control
  Interventions: Device: Allium ureteral stent

INTERVENTIONS:
Device: Allium ureteral stent — observe the effficacy and safety of long-term self expanding ureteral stents for treating refractory ureteral stricture

SUMMARY:
To conduct a prospective, multi-center study to observe the long-term efficacy and safety of self expanding ureteral stent for treating participants with refractory ureteral stricture.

DETAILED DESCRIPTION:
The aim of the study is to conduct a prospective, multi-center study to observe the long-term efficacy and safety of self expanding ureteral stent for treating participants with refractory ureteral stricture.

About 200 participants with refractory ureteral stricture will be enrolled in four hospitals. After the allium ureteral stents are placed, renal function, renal echo, images and associated complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* refractory ureteral stricture after at least two times of ureteral dilation

Exclusion Criteria:

* poor cardiovascular function for anesthesia unwilling to accept the long-term placement of ureteral stent uncontrolled urinary tract infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Renal function test | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months, 48 months, 54 months and 60 months
  serum creatinine (mg/dL)

SECONDARY OUTCOMES:
Complications | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months, 48 months, 54 months and 60 months
  device associated complications (e.g. urinary tract infection, stone formation, hematuria, stent migration)
Renal structure | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months, 48 months, 54 months and 60 months
  Renal echo (e.g. no hydronephrosis, mild hydronephrosis, moderate hydronephrosis, orsevere hydronephrosis)

CONTACTS AND LOCATIONS:
Overall Officials: Chung Cheng Wang, MD PhD, Principal Investigator — En Chu Kong Hospital
Locations (1):
- En Chu Kong Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Other researchers can e-mail to us for data sharing

REFERENCES:
- [Result] Avitan O, Bahouth Z, Shprits S, Gorenberg M, Halachmi S. Allium Ureteral Stent as a Treatment for Ureteral Stricture: Results and Concerns. Urol Int. 2022;106(5):482-486. doi: 10.1159/000522174. Epub 2022 Mar 1. PMID 35231922
- [Result] Sampogna G, Grasso A, Montanari E. Expandable metallic ureteral stent: indications and results. Minerva Urol Nefrol. 2018 Jun;70(3):275-285. doi: 10.23736/S0393-2249.18.03035-7. Epub 2018 Mar 28. PMID 29595037